CLINICAL TRIAL: NCT06719661
Title: The Impact of Clinical Pharmacist Intervention and Dapagliflozin as Add-On Therapy in the Management of Type 2 Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Mohammed Abdalaziz Hama amin, Principal Investigator, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH141-24
Record Dates: First submitted 2024-11-30; First posted 2024-12-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Uncontrolled type 2 diabetes; Dapagliflozin; Effects on HbA1c; Effects on body weight; Effects on fasting plasma glucose level
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dapagliflozin as add on therapy group (Experimental): Patients with uncontrolled type 2 diabetes receive dapagliflozin 10 mg once daily for 3 months as add-on therapy to their dual or triple standard therapy without receiving clinical pharmacist-led intervention.
  Interventions: Drug: Dapagliflozin 10mg
- Clinical pharmacist-led intervention group (Experimental): Patients with uncontrolled type 2 diabetes receive clinical pharmacist-led intervention, including dosage adjustment, dietary modification, education on the importance of adherence, strategies to improve adherence, and regular follow-up along with their standard dual or triple oral hypoglycemic medicines
  Interventions: Other: Clinical Pharmacist-led Intervention
- Standard therapy group (Other): Patients with uncontrolled type 2 diabetes receiving their standard dual or triple therapy only
  Interventions: Other: Standard therapy group

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Uncontrolled type 2 diabetic patients receive dapagliflozin 10 mg tablet once daily. They are asked to take it for 3 months, then return for their final assessment after 3 months
  Arms: Dapagliflozin as add on therapy group
Other: Clinical Pharmacist-led Intervention — Patients with uncontrolled type 2 diabetes will undergo dosage intensification of their dual or triple oral hypoglycemic medicines up to maximum daily doses. Further, they will be advised on specific dietary modification, education on the importance of adherence, strategies to improve adherence, including giving pill boxes, and regular follow-up every month via telephone-based communication.
  Arms: Clinical pharmacist-led intervention group
Other: Standard therapy group — Patients are receiving their standard dual or triple oral hypoglycemic therapy only.
  Arms: Standard therapy group

SUMMARY:
Diabetes mellitus is a progressive endocrine disease characterized by insulin deficiency with or without insulin resistance. Management of type 2 diabetes requires a comprehensive team following and monitoring the disease carefully. Dapagliflozin is a sodium-glucose co-transporter-2 (SGLT2) inhibitor, has been shown to be an effective medication for the treatment of T2DM, and has been demonstrated to improve glycemic control. The investigators believe that enrolling clinical pharmacist intervention as a part of a multidisciplinary approach and dapagliflozin is necessary to provide better patient care in patients that are on dual or triple oral hypoglycemic agents other than dapagliflozin. Therefore, the hypothesis of this study is that the impact and tolerability of clinical pharmacist-led intervention can be comparable to add on dapagliflozin alone on glycemic control in the management of T2DM.

DETAILED DESCRIPTION:
The study will be a three-arm prospective, randomized, controlled trial conducted in the Diabetes and endocrine center in Sulaymaniyah, Iraq. Participants will be randomly assigned to one of the following three groups. Group 1 receives dapagliflozin 10 mg as add-on therapy along with their standard dual or triple oral hypoglycemic medicines; group 2 receives clinical pharmacist-led intervention including dosage adjustment, dietary modification, education on the importance of adherence, strategies to improve adherence, and regular follow-up along with their standard dual or triple oral hypoglycemic medicines; group 3 is the standard therapy group when patients are receiving their standard dual or triple therapy only; and the duration of the study is 3 months. Glycemic control will be measured by measurement of HbA1c and fasting plasma glucose level after 3 months. Changes in body weight and BMI will also be done; in addition, compliance will be measured using a hill-bone compliance scale for high blood pressure medication applied to diabetic medication. The expected outcome includes improving both HbA1c and fasting plasma glucose levels in both groups compared to baseline and comparable improvement in parameters between the clinical pharmacist-led intervention group and dapagliflozin 10 mg add-on therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of type 2 diabetes mellitus having either dual or triple therapy, including (metformin, sulfonylurea, and/or DPP-4 inhibitors).
* HbA1c level between 7.0% and 10% and patients with HbA1c above 10% but refusing insulin therapy.
* Willing to provide informed consent.

Exclusion Criteria:

* Presence of comorbidities (e.g., severe renal impairment (eGFR < 30 mL/min/1.73m²), thyroid dysfunction, liver dysfunction).
* Presence of type 1 diabetes mellitus.
* History of diabetic ketoacidosis.
* Pregnancy or breastfeeding.
* Cognitive impairment or inability to provide informed consent.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months
  This measures changes in HbA1c from baseline to the end of the study period.
Fasting Plasma Glucose Level | 3 months
  This measures changes in fasting plasma glucose level from baseline to the end of the study period.
Body mass index (BMI) | 3 months
  This measures changes in weight in kg and height in meters to calculate changes of BMI (kg/m2) from baseline to the end of the study period.
Waist circumference | 3 months
  This measures changes in waist circumference in centimeters from baseline to the end of the study period.
Incidence of adverse events | 3 months
  This measures the reported incidence of adverse events, including urinary tract and genital infections and hypoglycemia.

SECONDARY OUTCOMES:
Modified Hill-bone compliance scale | 3 months
  This measures the difference in adherence of patients to their medicines between baseline and the end of the study period. The questionnaire is composed of 14 item questions: appointment-keeping questions (3-items), diet (2-items), and medication adherence (9-items). The response to each question is one of the following:
  1. All of the Time (Four marks)
  2. Most of the Time (Three marks)
  3. Some of the Time (Two Marks)
  4. None of the Time (One Mark) The interpretation of the scale is done based on the following: Patients with mark scores of 14-28 will be considered as having good or high compliance, and those with mark scores of 29-42 will be considered as having average or medium compliance, while those having mark scores of 43-56 will be considered as having poor or low compliance.
Lipid Profile | 3 months
  This measures changes in lipid profile (Total cholesterol, LDL, HDL and Triglyceride) from baseline to the end of the study period
Blood pressure | 3 months
  This measures changes in blood pressure from baseline to the end of the study period
Serum creatinine | 3 months
  This measures changes in serum creatinine from baseline to the end of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. Hama amin, BSc. Pharmacy, Principal Investigator — University of Sulaimani, College of Pharmacy; Rawa A. Ratha, Ph.D. Clinical Pharmacy, Principal Investigator — University of Sulaimani, College of Pharmacy; Taha O. Asaad, Professor, Principal Investigator — College of Medicine - University of Sulaimani
Locations (2):
- Iraq (2):
  - Endocrine and Diabetes Center, Sulaymaniyah, Kurdistan Region
  - Ministry of Higher Education and Scientific research, University of Sulaimani, College of Pharmacy, Sulaymaniyah, Kurdistan Region